CLINICAL TRIAL: NCT04586205
Title: A Pilot Proof of Concept, Within Subjects, Randomized Study of the Effects of Activation of the DLPFC Promotion System on TMS Treatment
Brief Title: Task Augmentation of Transcranial Magnetic Stimulation (TMS)
Acronym: TaskTMS
Status: Completed | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Yvette Sheline, Director, Center for Neuromodulation in Depression and Stress (CNDS), University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 832232
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: TMS; fMRI; dlPFC

STUDY DESIGN:
Intervention Model Description: A within-subjects design was used. Healthy participants between the ages of 18 and 60 who met basic eligibility criteria were invited to participate.
  In the first phase, all participants completed both the Sternberg task (SST) and the International Affective Picture System (IASP) task, each containing high- and low-load trials.
  In the second phase, participants completed the IASP task during two separate TMS sessions: one with active rTMS and one with sham rTMS, in a randomized crossover design. No TMS-alone condition was included. All TMS sessions were conducted in the MRI scanner, allowing investigators to collect both brain activation to single-pulse TMS probes and connectivity data.
  Participants were randomized to receive either active or sham rTMS during the first session, and then crossed over to the alternate condition after a two-week break. This design allowed for within-subject comparison of cortical response during the same task across both stimulation conditions.
Who Masked: Participant, Investigator
Oversight: Unapproved Device: Yes

ARMS (2):
- Active rTMS + IASP (Active Comparator): Participants perform the IASP emotional task Receive active rTMS
  Interventions: Device: active TMS; Behavioral: IASP Task; Behavioral: SST Task; Other: MRI
- Sham rTMS + IASP (Sham Comparator): Participants perform the IASP emotional task Receive Sham rTMS
  Interventions: Device: sham TMS; Behavioral: IASP Task; Behavioral: SST Task; Other: MRI

INTERVENTIONS:
Device: active TMS — Participants receive active repetitive transcranial magnetic stimulation (rTMS) while performing the International Affective Picture System (IASP). Stimulation is delivered at 120% of resting motor threshold (RMT), in triplet 50 Hz bursts, repeated at 5 Hz (2s on, 8s off), totaling 600 pulses per session.
  Arms: Active rTMS + IASP
Device: sham TMS — Participants receive sham rTMS while performing the IASP task. Stimulation is mimicked without actual neural activation using the same schedule and coil placement as the active condition.
  Arms: Sham rTMS + IASP
Behavioral: IASP Task — Participants complete the IASP (emotional image viewing) task during each TMS session (active and sham). The task includes both high- and low-load trials, designed to activate the dorsolateral prefrontal cortex (DLPFC). Task order and load levels are consistent across both stimulation sessions.
Behavioral: SST Task — In a separate MRI session prior to TMS sessions, participants complete the SST which includes both high-load and low-load trials. This cognitive task is used to examine baseline DLPFC activation and to contrast cognitive vs. emotional activation profiles.
Other: MRI — Participants undergo MRI sessions to measure DLPFC cortical reactivity and connectivity.

SUMMARY:
This pilot, within-subjects, randomized proof-of-concept study investigates the effects of activating the DLPFC promotion system on TMS treatment outcomes. Twenty-five healthy volunteers will participate in four sessions involving either active or sham repetitive transcranial magnetic stimulation (rTMS). Using anatomically guided TMS paired with cognitive tasks, the study tests the hypothesis that cognitive paired associative stimulation enhances cortical responses. For this pilot study, we are focusing only on the augmentation of TMS with the IASP task.

DETAILED DESCRIPTION:
The standard clinical use of repetitive transcranial magnetic stimulation (rTMS) for major depressive disorder (MDD) has shown limited efficacy. One contributing factor may be the common use of scalp-based targeting rather than neuronavigation techniques using functional MRI (fMRI), which enable more precise, individualized targeting of functional brain networks. Image-guided TMS can account for anatomical variability and may enhance treatment outcomes.

Another promising approach is combining TMS with concurrent cognitive activation of the dorsolateral prefrontal cortex (DLPFC). This concept, known as cognitive paired associative stimulation, builds on traditional paired associative stimulation (PAS), where coordinated stimulation enhances cortical response. In this framework, delivering TMS to the DLPFC while participants engage in a DLPFC-activating cognitive task could produce greater neural activation than either stimulus alone. Prior research suggests that the brain's cognitive or emotional state during stimulation can significantly modulate TMS effects, though it's unclear whether this enhancement depends on the type of cognitive task or the magnitude of neural activation.

Study Design and Procedure This within-subjects, mechanism-focused pilot study builds on the Research Domain Criteria (RDoC) framework for cognitive control. The primary goal is to examine how pairing rTMS with specific task conditions affects DLPFC activation and connectivity.

Participants (ages 18-60, healthy volunteers) will undergo the following:

Screening Visit (2 hours): Consent and eligibility. Visit 1 - Baseline MRI (1 hour): Participants undergo structural and functional MRI to localize the "Fitzgerald target" in the DLPFC. Data will be analyzed using FSL and neuronavigated using BrainSight.

Visit 2 - Task-Only fMRI Session (2 hours): Participants complete both the SST (cognitive task) and the IASP (emotional task) in the scanner. Each task contains high- and low-load trials, and participants complete both tasks (they are not assigned to one or the other).

Visits 3 & 4 - TMS Sessions (2 hours each): In a randomized crossover design, participants complete the IASP task while receiving either:

Active rTMS Sham rTMS These sessions test whether pairing emotional cognitive activation with TMS enhances cortical response. Note: TMS was never delivered alone-participants always performed the IASP task during stimulation.

2-Week Break Visits 5 & 6 - Follow-Up TMS Sessions (2 hours each): Participants repeat the IASP task with the alternate stimulation condition (sham or active). fMRI data is again collected to assess DLPFC activation and connectivity post-stimulation.

Each TMS session uses:

Stimulation Parameters: 120% resting motor threshold (RMT), triplet 50 Hz bursts at 5 Hz, 2s on / 8s off, 600 pulses per session (~3 min 9 sec total).

Probe Scans: Single-pulse TMS (120% RMT; 77 pulses/session) inside the scanner to measure cortical reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Gender, inclusive
* 18 60 years of age
* Right-handed
* No history of meeting Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria for any diagnosis
* Normal cognition
* Patients must be able to read and understand English
* Participants must be able to provide consent

Exclusion Criteria:

* Pregnancy (Female participants)
* Outside age range
* Meets DSM criteria for any diagnosis
* Unable to have an MRI scan
* Medical condition that interferes with the collection or interpretation of MRI data
* Implanted devices such as: aneurysm clip or cardiac pacemaker
* History of stroke, epilepsy, or brain scarring
* Cognitive impairment
* Recent use of psychoactive medications, as determined by investigators
* Otherwise determined by investigator to be unfit for participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-07 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2024-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuromodulation in Depression and Stress, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were a total of 17 people consented and completed the SST and emotion task during baseline (Week 1), three people withdrew, only 14 people completed the study,
  Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
Groups:
- Active Then Sham TMS Randomized: Of the 17 Participants to receive active TMS, 8 participants were randomized to active TMS first then received sham TMS after 2 week washout.
- Sham TMS vs Active TMS Randomised: Of the 17 Participants to receive active TMS, 9 participants were randomized to sham TMS first then received active TMS after 2 week washout.
Period: Baseline With MRI Scan, and SST and IAPS
Arm/Group | Active Then Sham TMS Randomized | Sham TMS vs Active TMS Randomised
Started (Each participant was took part in each arm of the study. There was a total of 17 people that consented, three people withdrew so only 14 people completed the study,) | 8 | 9
Active Then Sham TMS (8 participants were randomized to active TMS first then received sham TMS after 2 week washout. on withdrew from the study after the randomization.) | 8 | 0
Sham Then TMS (9 participants were randomized to sham TMS first then received active TMS after 2 week washout. 2 participants were withdrew from the study after the randomization.) | 0 | 9
Completed (Each participant was took part in each arm of the study. There was a total of 17 people that consented, three people withdrew so only 14 people completed the study.) | 7 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: TMS/Sham Visit, With IAPS
Arm/Group | Active Then Sham TMS Randomized | Sham TMS vs Active TMS Randomised
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Sham/TMS Visit, With IAPS
Arm/Group | Active Then Sham TMS Randomized | Sham TMS vs Active TMS Randomised
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: MRI Follow-Up
Arm/Group | Active Then Sham TMS Randomized | Sham TMS vs Active TMS Randomised
Started | 7 | 7
Completed (Each participant was took part in each arm of the study. There was a total of 17 people that consented, three people withdrew so only 14 people completed the study.) | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each participant was took part in each arm of the study. There was a total of 17 people that consented, three people withdrew so only 14 people completed the study,
Groups:
- Low-load Condition vs High-load: Participants will be assigned to complete either a high-load or a low-load cognition task. They will assigned to for both Sternberg task and emotional task.
  Sternberg Task: Participants will be randomized to high-load and low-load cognition task in different orders
- TMS vs. Task Order Completion: Participants will will then complete again (in randomized order) with rTMS:
  1. rTMS alone
  2. rTMS + SST (cognitive)
  3. rTMS + IAPS (emotion)
  Order of MRI procedures: Participants will be assigned to complete MRI+task, MRI +SST, and MRI + IAPS in random order
- Determination of Neuromodulation Effect on DLPFC Activation - Cognitive vs. Emotional: Participants will be assigned for the rest of the study to either complete their neuromodulation sessions while either completing the cognitive task, or the emotional task.
  TMS/Sham TMS: Participants will be randomized to either complete their assigned task (cognitive vs. emotional) while doing sham rTMS vs. real rTMS during weeks 2 and 3 of the study. The order of sham rTMS vs. real rTMS is randomized.
- Total: Total of all reporting groups
Arm/Group | Low-load Condition vs High-load | TMS vs. Task Order Completion | Determination of Neuromodulation Effect on DLPFC Activation - Cognitive vs. Emotional | Total
Number analyzed (Participants) | 17 | 0 | 0 | 17
Age, Categorical [Count of Participants; unit: Participants] — Each participant was took part in each arm of the study. There was a total of 17 people that consented, three people withdrew so only 14 people completed the study,
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 17 | 0 | 0 | 17
    >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (11.25) |  |  | 34 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 |  |  | 9
  Male | 8 |  |  | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 4 |  |  | 4
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 2 |  |  | 2
  White | 11 |  |  | 11
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 |  |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Sternberg Sorting Task (SST) at Baseline
Description: This Sternberg Sorting Task (SST) task is designed to assess how individuals store and retrieve random information from short-term memory. This task was administered to all participants before they were randomized into one of two groups (active TMS first then sham TMS or sham TMS first then active TMS). 0's were recorded for incorrect responses and 1's were recorded for correct responses. Therefore, the mean represents the accuracy percentage for each group.
Time Frame: Baseline (Visit 1)
Population: There were a total of 17 people that consented, one person that was receiving active TMS first withdrew from the study and two people that were receiving sham TMS first withdrew from the study so only 14 people completed. (seven receiving Active TMS first and seven that were receiving sham TMS first).
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Groups:
- Baseline Measurement Before Active TMS vs Sham TMS: Participants that were randomized to active TMS first then received sham TMS after 2 week washout
- Baseline Measurement Before Sham TMS vs Active TMS: Participants that were randomized to sham TMS first then received active TMS after 2 week washout
Arm/Group | Baseline Measurement Before Active TMS vs Sham TMS | Baseline Measurement Before Sham TMS vs Active TMS
Number analyzed (Participants) | 8 | 9
proportion of correct responses
  High-Load SST | 0.85 (0.17) | 0.64 (0.31)
  Low-Load SST | 0.87 (0.065) | 0.66 (0.34)
Statistical Analysis 1: Comparison: Baseline Measurement Before Active TMS vs Sham TMS; The baseline measurement for this analysis is the Sternberg Sorting Task (SST) at Baseline. This task is designed to assess how individuals store and retrieve random information from short-term memory. This task was administered to all participants before they were randomized into one of two groups (active TMS first then sham TMS or sham TMS first then active TMS); Test type: Other; p = 0.024, ANOVA

2. Primary Outcome: International Affective Picture System (IAPS)
Description: International Affective Picture System (IAPS): an emotional task using IAPS picture that will also compare low load and high load conditions. The number of images will vary by condition load, but for both the high-load & low-load conditions, participants will look at IAPS pictures and answer questions about the images. Further, jittered within this design will be both neutral and negative blocks of IAPS pictures: Baseline measurement before randomizing participants into Active or Sham groups. 0's were recorded for incorrect responses and 1's were recorded for correct responses. Therefore, the mean represents the accuracy percentage for each group.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of correct responses
Groups:
- Baseline Measurement Before Active vs Sham TMS: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
  Participants will be randomized to receive either sham TMS first and then active TMS, or active TMS and then sham TMS.
- Baseline Measurement Before Sham TMS Then Active TMS: 9 participants were randomized to sham TMS first then received active TMS after 2 week washout
Arm/Group | Baseline Measurement Before Active vs Sham TMS | Baseline Measurement Before Sham TMS Then Active TMS
Number analyzed (Participants) | 8 | 9
proportion of correct responses
  High-Load IAPS | 0.69 (0.21) | 0.52 (0.14)
  Low-Load IAPS | 0.67 (0.09) | 0.59 (0.22)
Statistical Analysis 1: Comparison: Baseline Measurement Before Active vs Sham TMS; The baseline measurement for this analysis is the International Affective Picture System (IAPS) at baseline. This is an emotional task using IAPS picture that will also compare low load and high load conditions. The number of images will vary by condition load, but for both the high-load & low-load conditions, participants will look at IAPS pictures and answer questions about the images. We compare mean High-Load IAPS and Low-Load IAPS scores in the group that received active then sham TMS; Test type: Other; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = .02 — The difference in means between High-Load IAPS (.69) and Low-Load IAPS (.67) in the group that received active then sham TMS

3. Secondary Outcome: International Affective Picture System (IAPS) at Post-intervention (Active/Sham)
Description: These measurements were taken at the final visits. For example, the "Active then Sham TMS" group received sham TMS during this outcome measure, and the opposite for "Sham then Active TMS." International Affective Picture System (IAPS): an emotional task using IAPS picture that will also compare low load and high load conditions. The number of images will vary by condition load, but for both the high-load & low-load conditions, participants will look at IAPS pictures and answer questions about the images. Further, jittered within this design will be both neutral and negative blocks of IAPS pictures. The mean represents the number of correct responses from each group. Values can range from 0-299 for the High-Load IAPS (0 meaning no answers correct, and 299 meaning all answers correct). Values can range from 0-326 for the Low-Load IAPS (0 meaning no answers correct, and 326 meaning all answers correct).
Time Frame: post-intervention (Active/Sham) (Week 6 Final Visit)
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Active Then Sham TMS: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
  This group is for participants that were randomized to receive active TMS, and then received sham TMS after a two week washout period.
  Since this outcome variable is for the final visits, this group received Sham TMS for this measure.
- Sham Then Active TMS: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
  This group is for participants that were randomized to receive sham TMS, and then received active TMS after a two week washout period.
  Since this outcome variable is for the final visits, this group received Active TMS for this measure.
Arm/Group | Active Then Sham TMS | Sham Then Active TMS
Number analyzed (Participants) | 7 | 7
units on a scale
  High-Load IAPS | 178 [0 to 299] | 121 [0 to 299]
  Low-Load IAPS | 193 [0 to 326] | 223 [0 to 326]
Statistical Analysis 1: Comparison: Active Then Sham TMS; The outcome measure for this analysis was the International Affective Picture System (IAPS); Test type: Other; p = 0.19, Chi-squared

4. Secondary Outcome: Comparing the Impact of Sternberg Sort Task (SST), the Working Memory Task and International Affective Picture System (IAPS) Emotional Task on TMS-Induced DLPFC Activation; Post-intervention (Active/Sham)
Description: In the final visit, we recorded these following tasks in an MRI, in both the group that received active then sham TMS and the group that received sham then active TMS. We are comparing the effects of two distinct cognitive tasks on augmenting the impact of TMS on dorsolateral prefrontal cortex (DLPFC) activity. The first task is the Sternberg task (SST), a working memory task designed to engage cognitive processes by requiring participants to retain and recall information. The second is the International Affective Picture System (IAPS) task, which presents emotionally evocative images to elicit emotional responses. Our goal is to determine which task-cognitive or emotional-more effectively enhances TMS-induced DLPFC activation. Brain activity and connectivity can be quantified on a normalized scale ranging from 0 to 1, where 0 indicates no detectable activity or connectivity, and 1 represents the highest level of activity or connectivity within the measured range.
Time Frame: post-intervention (Active/Sham) (Week 6 Final Visit)
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Active Then Sham TMS: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
  This group is for participants that were randomized to receive active TMS, and then received sham TMS after a two week washout period.
- Sham Then Active TMS: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first. All participants that completed the study, completed the emotional IAPS task high load and low load.
  This group is for participants that were randomized to receive sham TMS, and then received active TMS after a two week washout period.
Arm/Group | Active Then Sham TMS | Sham Then Active TMS
Number analyzed (Participants) | 7 | 7
score on a scale
  High-Load SST | 0.266 [0 to 1] | 0.183 [0 to 1]
  Low-Load SST | 0.156 [0 to 1] | 0.056 [0 to 1]
  High-Load IAPS | 0.232 [0 to 1] | 0.135 [0 to 1]
  Low-Load IAPS | 0.201 [0 to 1] | 0.129 [0 to 1]
Statistical Analysis 1: Comparison: Active Then Sham TMS; Test type: Superiority; p = 0.67, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Description: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first.
  Each participant completed a Baseline visit before being randomized, and all adverse events were recorded from the time the participant signed the consent form until study completion.
  Adverse events were reported as 2 groups: The group that received active then sham, and the group that received sham then active.
Groups:
- Active TMS Then Sham TMS Group: MRI; Active TMS Then Sham TMS Group: Active TMS; Active TMS Then Sham TMS Group: Sham TMS; Active TMS Then Sham TMS Group: SST Task; Active TMS Then Sham TMS Group: IASP Task: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first.
  8 participants were randomized to active TMS first then received sham TMS after 2 week washout.
  Each participant completed a Baseline visit before being randomized, and all adverse events were recorded from the time the participant signed the consent form until study completion.
  One participant in this group experienced mild pain in the head during the TMS intervention period.
- Sham TMS Then Active TMS: MRI; Sham TMS Then Active TMS: Active TMS; Sham TMS Then Active TMS: Sham TMS; Sham TMS Then Active TMS: SST Task; Sham TMS Then Active TMS: IASP Task: Each participant took part in both sham TMS and active TMS. They were randomized into which treatment they would receive first.
  9 participants were randomized to sham TMS first then received active TMS after 2 week washout.
  Each participant completed a Baseline visit before being randomized, and all adverse events were recorded from the time the participant signed the consent form until study completion.
Arm/Group | Active TMS Then Sham TMS Group: MRI | Sham TMS Then Active TMS: MRI | Active TMS Then Sham TMS Group: Active TMS | Sham TMS Then Active TMS: Active TMS | Active TMS Then Sham TMS Group: Sham TMS | Sham TMS Then Active TMS: Sham TMS | Active TMS Then Sham TMS Group: SST Task | Sham TMS Then Active TMS: SST Task | Active TMS Then Sham TMS Group: IASP Task | Sham TMS Then Active TMS: IASP Task
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 1/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9 | 0/8 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS Then Sham TMS Group: MRI (N=8) | Sham TMS Then Active TMS: MRI (N=9) | Active TMS Then Sham TMS Group: Active TMS (N=8) | Sham TMS Then Active TMS: Active TMS (N=9) | Active TMS Then Sham TMS Group: Sham TMS (N=8) | Sham TMS Then Active TMS: Sham TMS (N=9) | Active TMS Then Sham TMS Group: SST Task (N=8) | Sham TMS Then Active TMS: SST Task (N=9) | Active TMS Then Sham TMS Group: IASP Task (N=8) | Sham TMS Then Active TMS: IASP Task (N=9)
Mild Pain in Head (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT04586205/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT04586205/ICF_001.pdf